CLINICAL TRIAL: NCT02406261
Title: A Study to Characterize LY3314814 Pharmacokinetics as a Function of Dosing Duration and to Determine the Effect of LY3314814 on the Pharmacokinetics of CYP3A Substrates in Healthy Subjects
Brief Title: A Drug-Drug Interaction Study of Lanabecestat (LY3314814) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16014; I8D-MC-AZER (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-02; First posted 2015-04-02 (Estimated); Results first posted 2019-03-22 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — lanabecestat; Simvastatin; Midazolam; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort A (Experimental): 500 microgram (mcg) midazolam, single oral dose on Days 1, 17, and 35;
  20 mg simvastatin, single oral dose on Days 2 and 36;
  250 microgram (mcg) midazolam, intravenous (IV) on Days 3 and 37;
  50 mg lanabecestat, single oral dose on Day 4;
  50 mg lanabecestat, single oral dose, Days 10 to 37
  Interventions: Drug: Lanabecestat; Drug: Simvastatin; Drug: Midazolam
- Cohort B (Experimental): 5 mg donepezil, single oral dose on Day 1, Period 1;
  50 mg lanabecestat, single oral dose Days 1 to 43, Period 2;
  5 mg donepezil, single oral dose on Day 28, Period 2
  Interventions: Drug: Donepezil; Drug: Lanabecestat

INTERVENTIONS:
Drug: Lanabecestat — 50 mg lanabecestat will be administered orally as 1 × 50-mg tablet
  Other Names: LY3314814; AZD3293
  Arms: Cohort A
Drug: Simvastatin — 20 mg simvastatin will be administered orally as 1 × 20-mg tablet
  Arms: Cohort A
Drug: Midazolam — 500 mcg midazolam will be administered orally as 0.25 mL of 2-mg/mL syrup
  Arms: Cohort A
Drug: Midazolam — 250 mcg midazolam will be administered intravenous (IV) as 0.25 mL of 1-mg/mL injection solution
  Arms: Cohort A
Drug: Donepezil — 5 mg donepezil will be administered orally as 1 × 5-mg tablet
  Arms: Cohort B
Drug: Lanabecestat — 50 mg lanabecestat will be administered orally as 1 × 50-mg tablet
  Other Names: LY3314814; AZD3293
  Arms: Cohort B

SUMMARY:
The purpose of this study is to study the effect of lanabecestat on how the body absorbs and processes 3 other medications, midazolam, simvastatin and donepezil and how these 3 medications affect lanabecestat when they are taken together. This study is in 2 cohorts, Cohort A is approximately 44 days long and Cohort B about 70 days only. The screening visit is required within 30 days prior to the start on the study

DETAILED DESCRIPTION:
Astra Zeneca (AZ) registered this trial as sponsor. In July, 2015, sponsorship changed to Eli Lilly and Company (Lilly). In August, 2015, AZ transferred this trial to Lilly's ClinicalTrials.gov account and Lilly updated the record. This trial is not an applicable trial under the Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy and either sterile or, male and prepared to use an approved method of contraception
* Have a body mass index (BMI) at screening of 19.0 to 32.0 kilogram per square meter (kg/m^2)

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may put the subject at risk because of participation in the study, may influence the results, or may limit the subject's ability to participate in the study
* History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
* History of previous or ongoing psychiatric disease/condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2015-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Covance Inc, Daytona Beach, Florida
  - Covance Inc, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned that all subjects in Cohort B would be enrolled at Site 002.
Groups:
- Cohort A: 500 microgram (mcg) midazolam, single oral dose on Days 1, 17, and 35; 20 mg simvastatin, single oral dose on Days 2 and 36; 250 mcg midazolam, intravenous (IV) on Days 3 and 37; 50 mg LY3314814, single oral dose on Day 4; 50 mg LY3314814, single oral dose, Days 10 to 37
- Cohort B: 5 mg donepezil, single oral dose on Day 1 Period 1; 50 mg LY3314814, single oral dose Days 1 to 43, Period 2; 5 mg donepezil, single oral dose on Day 28 Period 2
Period: Period 1
Arm/Group | Cohort A | Cohort B
Started | 50 | 32
Received at Least One Dose of Study Drug | 50 | 32
Completed | 47 | 32
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Adverse Event | 1 | 0
Period: Period 2
Arm/Group | Cohort A | Cohort B
Started | 0 (Cohort A participated in Period 1 only) | 32
Completed | 0 | 29
Not Completed | 0 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: 500 microgram (mcg) midazolam, single oral dose on Days 1, 17, and 35; 20 mg simvastatin, single oral dose on Days 2 and 36; 250 microgram (mcg) midazolam, intravenous (IV) on Days 3 and 37; 50 mg LY3314814, single oral dose on Day 4; 50 mg LY3314814, single oral dose, Days 10 to 37
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Total
Number analyzed (Participants) | 50 | 32 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 32 | 82
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 26
  Male | 34 | 22 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 7 | 28
  Not Hispanic or Latino | 29 | 25 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 14 | 34
  White | 27 | 16 | 43
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 32 | 82

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK): Area Under the Curve Zero to Infinity (AUC[0-∞]) for LY3314814
Time Frame: Day 4: Predose, 0.5, 1, 2, 3, 4, 8, 12, 24, 48, 72, 96, and 120 hours (Cohort A)
Population: Participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram * hour per milliliter (ng*h/mL)
Arm/Group | Cohort A
Number analyzed (Participants) | 50
Nanogram * hour per milliliter (ng*h/mL) | 3200 (21)

2. Primary Outcome: PK Profile for Simvastatin: AUC(0-∞)
Time Frame: Day 2 and 36: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours (Cohort A)
Population: Participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort A
Number analyzed (Participants) | 49
ng*h/mL
  AUC(0-∞) Simvastatin Day 2: number analyzed (Participants) | 44
  AUC(0-∞) Simvastatin Day 2 | 15.1 (84)
  AUC(0-∞) Simvastatin Day 36: number analyzed (Participants) | 48
  AUC(0-∞) Simvastatin Day 36 | 21.2 (59)

3. Primary Outcome: PK Profile for Midazolam: AUC(0-∞) Oral and IV Dose
Time Frame: Day 1, 3, 17, 35, and 37: Predose, 0.25, 0.5, 1, 2, 3, 5, 8, and 12 hours (Cohort A)
Population: Participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort A
Number analyzed (Participants) | 49
ng*h/mL
  AUC(0-∞) Oral Day 1 | 6.53 (38)
  AUC(0-∞) Oral Day 17 | 6.24 (42)
  AUC(0-∞) Oral Day 35 | 5.59 (40)
  AUC(0-∞) IV Day 3 | 11.4 (22)
  AUC(0-∞) IV Day 37: number analyzed (Participants) | 47
  AUC(0-∞) IV Day 37 | 11.6 (21)

4. Primary Outcome: PK Profile for Donepezil: AUC(0-∞)
Time Frame: Day 1 and 28: predose 0.5,1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96,120, 216, 288, and 360 hours (Cohort B)
Population: Participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort B
Number analyzed (Participants) | 31
ng*h/mL
  Day 1 | 271 (28)
  Day 28: number analyzed (Participants) | 29
  Day 28 | 285 (23)

5. Secondary Outcome: Number of Participants With One or More Serious Adverse Events(s) Considered by the Investigator to be Related to Study Drug Administration
Time Frame: Cohort A : Baseline to Study Completion (Up to Day 50); Cohort B: Baseline to Study Completion (Up to Day 70)
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 50 | 32
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Suicidal Ideation or Suicidal Behavior Based on Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS captures occurrence, severity, and frequency of suicide-related thoughts and behaviors. Suicidal behavior is defined as a "yes" answer to any of 5 suicidal behavior questions: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, and completed suicide. Suicidal ideation is defined as a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, and 4 different categories of active suicidal ideation.
Time Frame: Cohort A: Baseline to Study Completion (Up to Day 50); Cohort B: Baseline to Study Completion (Up to Day 70)
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A | Cohort B
Number analyzed (Participants) | 50 | 32
Participants
  Suicidal Ideation | 0 | 0
  Suicidal Behavior | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort A | Cohort B
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/32
Other Adverse Events (participants affected / at risk) | 6/50 | 7/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=50) | Cohort B (N=32)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days